CLINICAL TRIAL: NCT06714526
Title: Effect of Genotype-Guided Oral P2Y12 Inhibitor Selection vs Conventional Clopidogrel Therapy in Symptomatic Intracranial Atherosclerotic Disease: A Pilot Prospective, Randomized, Open-label, Blinded-endpoint (PROBE) Multi- Centre Study
Brief Title: Effect of Genotype-Guided Oral P2Y12 Inhibitor Selection vs Conventional Clopidogrel Therapy in Symptomatic ICAD
Acronym: NUANCE-ICAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5902
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Point-of-Care CYP2C19 Testing (Experimental): Patients will undergo point-of-care CYP2C19 testing with the Research Use Only (RUO) Genomadix Cube to inform the choice of P2Y12 inhibitor (i.e. clopidogrel vs ticagrelor).
  Interventions: Genetic: Point-of-Care CYP2C19 Testing; Drug: ticagrelor + aspirin; Drug: clopidogrel + aspirin
- Standard of Care (No Intervention): Patients will receive standard-of-care ASA + clopidogrel.

INTERVENTIONS:
Genetic: Point-of-Care CYP2C19 Testing — Genetic testing with the Genomadix cube to determine P2Y12 inhibitor
  Arms: Point-of-Care CYP2C19 Testing
Drug: ticagrelor + aspirin — If patients are poor or intermediate metabolizers of clopidogrel, they will receive ticagrelor (90 mg PO BID) + aspirin (81 mg PO daily)
  Arms: Point-of-Care CYP2C19 Testing
Drug: clopidogrel + aspirin — Normal, rapid, and ultra-rapid metabolizers of clopidogrel will receive 75 mg PO daily of clopidogrel and 81 mg PO daily of aspirin.
  Arms: Point-of-Care CYP2C19 Testing

SUMMARY:
Stroke is an important cause of death, disability, and memory problems in adults. The build-up of plaque in arteries inside the brain is known as "intracranial atherosclerotic disease" or "ICAD" for short, and can reduce blood flow in the brain. Clopidogrel is a medicine used to prevent strokes because it stops blood from clotting. However, there are some people who do not get as much benefit from Clopidogrel because of differences in their genes; they have a variation in a certain gene and their body is not able to properly process Clopidogrel. Another medication called Ticagrelor can benefit people who have this genetic variation. The study investigators will randomize patients who have had a stroke due to ICAD to receive genetic testing, or standard of care. The standard-of-care group will take Clopidogrel for 90 days. The genetic testing group will complete a genetic test to see if they can properly process Clopidogrel. Depending on the results of the genetic test, patients will either take Clopidogrel or Ticagrelor for 90 days. All patients will have a brain scan at baseline and 90 days to see if they had any new strokes. Patients will also complete tests and questionnaires about function and memory at baseline and 90 days. This study will be one of the first to see if it is feasible and safe to use genetic testing to help choose medications for patients who have had a stroke. This will help the study investigators design a larger study that can test if genetic testing in stroke patients reduces future stroke risk and improves health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years old, male and female.
* TIA or ischemic stroke secondary to symptomatic atherosclerotic stenosis of 30- 99% involving the intracranial ICA or MCA or posterior circulation arteries as evidenced by CT or MR angiography.
* Index TIA or ischemic stroke event occurred within past 30 days.
* Clinical indication for DAPT for at least 3 months.

Exclusion Criteria:

* Any contraindication to DAPT.
* Any contraindication to use of clopidogrel (Plavix) or ticagrelor (Brilinta), such as pregnancy. A pregnancy test will be performed on all women of child-bearing age prior to enrollment in the study.
* Indication for chronic anticoagulation based on guideline recommendations or investigator's judgment (e.g., atrial fibrillation, mechanical heart valve, intracardiac clot, dilated cardiomyopathy, ejection fraction <30%, etc.).
* Intracranial arterial occlusion (i.e. 100% stenosis) responsible for the acute brain ischemia.
* Intracranial arterial stenosis secondary to causes other than atherosclerosis.
* Extracranial carotid disease with a plan for carotid revascularization.
* Intraluminal thrombus.
* Unstable subdural hematoma within 12 months of randomization not amenable to embolization.
* Previous spontaneous hemorrhagic stroke.
* Traumatic brain hemorrhage within 1 month of randomization.
* Living in a nursing home or requiring daily nursing care or assistance with activities of daily living.
* Intracranial tumor (except meningioma) or any intracranial vascular malformation.
* Life expectancy less than 6 months.
* Enrolment in another study that would conflict with the current study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | Through study completion, an average of 90 days
  The number of patients who provide informed consent, or are deemed ineligible after screening.
Rate of study completion | Through study completion, an average of 90 days
  The number of patients who complete the entire study protocol
Rate of protocol deviations | Through study completion, an average of 90 days
  The number of patients who encounter at least one protocol deviation during the study
Proportion of patients with Symptomatic intracerebral hemorrhage (ICH) | Through study completion, an average of 90 days
  New symptomatic ICH OR worsening existing ICH with a ≥33% increase in hematoma volume AND NIHSS score increase of ≥4 points AND clinical change is thought to be attributable to ICH
Proportion of patients with major extracranial bleeding | Through study completion, an average of 90 days
  Bleeding in a critical area or organ, including intraspinal, intraocular, retroperitoneal, intra-articular, pericardial, intramuscular with compartment syndrome, and/or bleeding causing a drop in hemoglobulin by 20g/L or more
Proportion of patients with non-bleeding adverse events | Through study completion, an average of 90 days
  Non-bleeding adverse events related to the study drug including dyspnea, bradyarrhythmia, and/or chest pain

SECONDARY OUTCOMES:
Proportion of patients who have Microembolic Signals on Transcranial Doppler Ultrasound | Day 5 ± 2
Change in volume of ischemic strokes and white matter hyperintensities (optional) | Day 0 + 14 and Day 90 ± 14
Change in number of ischemic strokes and white matter hyperintensities | Day 0 + 3 and Day 90 ± 14
Number of patients with ischemic stroke, myocardial infarction, or death | Day 90 ± 14
Change in Montreal Cognitive Assessment (MoCA) score from baseline to follow-up | Day 0 and Day 90 ± 14
  To MoCA is a validated cognitive screening tool. Possible scores range from 0 (worst score) to 31 (best score). Change = Follow-up - baseline.
Change in NIH Stroke Scale (NIHSS) score from baseline to follow-up | Day 0 and Day 90 ± 14
  This scale is a 15 item tool used to quantify stroke severity. Scores range from 0 (no stroke) to 42 (most severe stroke). Change = Follow-up - baseline.
Change or shift in modified Rankin Scale (mRS) score from baseline to follow-up | Day 0 and Day 90 ± 14
  The MRS is a single item rating of stroke outcomes. Scores range from 0 (no symptoms) to 6 (death). Change = Follow-up - baseline.
Self-reported Quality of Life as assessed by the EQ-5D-5L | Day 90 ± 14
  The EQ-5D-5L questionnaire has 5 dimensions: Mobility, Self-Care, Usual Activity, Pain/Discomfort, Anxiety/Depression, with each dimension rated on a level from 1-5 where higher scores indicate more severe problems.
Self-reported Dementia Screening assessed by the AD8 Dementia Screening Interview | Day 90 ± 14
  The AD8 Dementia Screening Interview has 8 questions that ask if there has been a change in the last several years caused by cognitive (thinking and memory) problems. The score is the sum of all items marked "Yes, A change".
Self-reported functional status assessed by the Lawton-Brody Instrumental Activities of Daily Living Scale | Day 90 ± 14
  The Lawton-Brody Instrumental Activities of Daily Living Scale has 8 categories where participants can rate their functional level. Scores range from 0 (low function, dependent) to 8 (high function, independent).

CONTACTS AND LOCATIONS:
Overall Officials: Mark I Boulos, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Dr. Mark I. Boulos - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No